CLINICAL TRIAL: NCT07308197
Title: Effect of (Posterior Colpotomy First) Technique on the Vaginal Length During Total Abdominal Hysterectomy
Brief Title: Effect of Posterior Colpotomy First Technique on the Vaginal Length During Total Abdominal Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 367
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Hysterectomy, Benign Uterine Diseases
Keywords: hystrectomy; posterior colopotomy; Vaginal length

STUDY DESIGN:
Intervention Model Description: A lower midline or Pfannestiel incision is the first step in the complete abdominal hysterectomy procedure. They clamp, cut, and ligate the top pedicles. The cardinal and uterosacral ligaments were dissected, the wide ligament's leaves were cut, the bladder was carefully lowered, and the uterine vessels were skeletonized, cut, and tied.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Classic technique): (Active Comparator): the surgeon makes a circumferential incision after initially entering the front vaginal wall. The surgeon performs a circumferential colpotomy at the topmost section of the vagina
  Interventions: Procedure: Abdominal hysterectomy
- Group B (posterior colpotomy first) approach (Active Comparator): entering the vagina via the posterior wall at the uppermost part of the uterosacral ligaments, followed by the left lateral fornix
  Interventions: Procedure: Abdominal hysterectomy

INTERVENTIONS:
Procedure: Abdominal hysterectomy — A lower midline or Pfannestiel incision is the first step in the complete abdominal hysterectomy procedure. They clamp, cut, and ligate the top pedicles. The cardinal and uterosacral ligaments were dissected, the wide ligament's leaves were cut, the bladder was carefully lowered, and the uterine vessels were skeletonized, cut, and tied

SUMMARY:
the same surgeon performed all of the procedures using the same method. A lower midline or Pfannestiel incision is the first step in the complete abdominal hysterectomy procedure. They clamp, cut, and ligate the top pedicles. The cardinal and uterosacral ligaments were dissected, the wide ligament's leaves were cut, the bladder was carefully lowered, and the uterine vessels were skeletonized, cut, and tied. Group A (traditional technique): the surgeon makes a circumferential incision after initially entering the front vaginal wall. The surgeon performs a circumferential colpotomy at the topmost section of the vagina using the Group B (posterior colpotomy first) approach, entering the vagina via the posterior wall at the uppermost part of the uterosacral ligaments, followed by the left lateral fornix.

Reconstruction of the pelvic floor to ensure hemostasis and good pelvic support. The operative time was assessed by calculating the time between vaginal cuff opening and suturing after uterine artery ligation, As point D on the POP-Q system is omitted after hysterectomy, point C level was reassessed 2 weeks postoperative.

DETAILED DESCRIPTION:
the same surgeon performed all of the procedures using the same method. A lower midline or Pfannestiel incision is the first step in the complete abdominal hysterectomy procedure. They clamp, cut, and ligate the top pedicles. The cardinal and uterosacral ligaments were dissected, the wide ligament's leaves were cut, the bladder was carefully lowered, and the uterine vessels were skeletonized, cut, and tied. Group A (traditional technique): the surgeon makes a circumferential incision after initially entering the front vaginal wall. The surgeon performs a circumferential colpotomy at the topmost section of the vagina using the Group B (posterior colpotomy first) approach, entering the vagina via the posterior wall at the uppermost part of the uterosacral ligaments, followed by the left lateral fornix.

Reconstruction of the pelvic floor to ensure hemostasis and good pelvic support. The operative time was assessed by calculating the time between vaginal cuff opening and suturing after uterine artery ligation, As point D on the POP-Q system is omitted after hysterectomy, point C level was reassessed 2 weeks postoperative.

Total vaginal shortening (TVS) and vaginal shortening ratio (VSR) were calculated according to the formulas given below.

TVS=Preoperative VL-Postoperative VL at 3 months. VSP=Preoperative VL-Postoperative VL at 3 months\ Preoperative VL*100

ELIGIBILITY:
Inclusion Criteria:

* Ages 40 - 65 years
* sexually active
* BMI of 25-40 kg/m2
* had a fresh abdomen
* had a benign reason for a hysterectomy (multiple fibroid uterus, adenomyosis, or endometrial hyperplasia).

Exclusion Criteria:

* Patients who had vaginal and uterine prolapse,
* subtotal hysterectomy,
* caesarean hysterectomy in patients with major obstetric hemorrhage (placenta previa, accreta-increta-percreta, uncontrolled postpartum hemorrhage)
* malignant indications of total abdominal hysterectomy (uterine and cervical carcinoma)

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
Total vaginal length | after 3 months
  calculated according to the formula TVS=Preoperative VL-Postoperative VL

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — Cairo University
Locations (1):
- Cairo university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided